CLINICAL TRIAL: NCT04729504
Title: Cultural Adaptation and Dissemination of a Single-Session Intervention (SSI) Targeting Caregivers of Youth With Anxiety
Brief Title: Cultural Adaptation of a SSI for Youth Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jill May Ehrenreich, Professor, Department of Psychology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20210016
Record Dates: First submitted 2021-01-12; First posted 2021-01-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Project BRAVE Group (Other): Participants in this group will receive a single session intervention of a culturally and linguistically adapted Project BRAVE.
  Interventions: Behavioral: Adapted Project BRAVE

INTERVENTIONS:
Behavioral: Adapted Project BRAVE — A culturally and linguistically adapted Project BRAVE is web-based single session intervention that is about 30 minutes in length. The session is designed to focus on targeting child anxiety symptoms in the multilingual and diverse families in Miami-Dade.

SUMMARY:
The overarching objective of this protocol is to (1) adapt and (2) disseminate an evidence-based, brief (approximately 30 minute) single session intervention (SSI) to better reflect the cultural and linguistic diversity of Latin, Haitian, and Haitian-American individuals via a fully online platform.

ELIGIBILITY:
Inclusion Criteria:

1. Be caregivers (e.g. biological or adoptive parent, or legal guardian) of a child age 4-10.
2. Affirm that they have read the consent language and study overview on REDCap by checking a box.

Exclusion Criteria:

- Not meet all of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-12-21 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety as measured by GAD-2 | Baseline, 2 weeks
  Generalized Anxiety Disorder 2-item (GAD-2) Scale has a total score ranging from 0 to 6 with a score of 3 being the cut-off for identifying possible cases and in which further diagnostic evaluation for generalized anxiety disorder is warranted.
Change in anxiety as measured by the FASA | Baseline, 2 weeks
  Family Accommodation Scale - Anxiety (FASA) is a 9-item scale of measuring caregiver accommodation behaviors (modification of routines, facilitating avoidance, etc.) in light of youth anxiety. It has a total score ranging from 0 to 36 with the higher score indicating more frequent parental accommodation.
Program Feedback Scale (PFS) Scores | 2 weeks
  The PFS is a reliable, valid measure of the perceived acceptability of single-session interventions. It asks participants to rate acceptability and feasibility of an SSI they just completed. It has a total score ranging from 0 to 28 with the higher score indicating perceived acceptability and feasibility of the program.

SECONDARY OUTCOMES:
Perceived Change in Problem-Solving, and Preparedness to Manage Distress | 2 weeks
  Two questions (Schleider et al., 2020) will be used to assess change in ability to solve problems, and ability to manage distress. Participants will be asked, "to what extent are you able to solve the problems [with your child's anxiety] facing right now?", and "how prepared do you feel to manage [your child with] distressing situations?" It has a total score ranging from 2 to 10, with a higher score indicating better ability to solve problems, and to manage distress.
Change in State Hope Scale Scores | Baseline, 2 weeks
  State Hope Scale is a 6-item self-report scale designed to evaluate hope in adolescents and adults, including two reliable subscales: agency and pathways. It has a total score ranging from 6 to 48 with the higher scores representing higher hope levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ehrenreich-May, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No